CLINICAL TRIAL: NCT05867615
Title: Radiometabolic Therapy (RMT) With 177Lu PSMA in PSMA PET/CT Positive Advanced/Metastatic Tumours: a Basket Trial
Brief Title: Radiometabolic Therapy With 177Lu PSMA in PSMA PET/CT Positive Advanced/Metastatic Tumours:
Acronym: LUBASKET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST100.58
Record Dates: First submitted 2023-03-24; First posted 2023-05-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: basket study; PSMA PET/CT positive
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [177Lu]Lu-PSMA I&T (Experimental): [177Lu]Lu-PSMA I&T, intravenous, dosage of 5.5 - 7.4 GBq every 8 weeks
  Interventions: Drug: [177Lu]Lu-PSMA I&T

INTERVENTIONS:
Drug: [177Lu]Lu-PSMA I&T — 177Lu activity to be administered to single patient (range 5.5-7.4 GBq), every 8 weeks (±2 weeks) will be measured in a dose calibrator, properly calibrated for the radionuclide. The radiopharmaceutical will be slowly infused intravenously over 15-30' in a dedicated room using a dedicated pump system.

SUMMARY:
Phase 2 study, single arm trial enrolling patients with a Gallium-68/Fluorine-18 prostate-specific membrane antigen (PSMA) positive positron emission tomography/Computed Tomography (PET/CT) in order to be treated with Lutetium-177 (177Lu) PSMA.

Patients without risk factors for toxicity will receive 7.4 GBq of 177Lu-PSMA while patients with at least 1 risk factor for toxicity will receive 5.5 GBq of 177Lu-PSMA. Patients will receive 4 cycles every 8 weeks (+- 2 weeks)

DETAILED DESCRIPTION:
Since PSMA radioligand therapy (PSMA-RLT) demonstrated remarkable therapeutic efficacy in prostate cancer patients, the question arises whether PSMA-RLT could also achieve beneficial effects in other cancers expressing PSMA on the tumors cells themselves, or in the tumor-associated neovasculature. Expression of PSMA was early-on also identified in kidney, salivary glands, the duodenum and the central and peripheral nervous system. Subsequently, a wide variety of immunohistochemistry (IHC) studies showed PSMA to be upregulated on the endothelial cells of the neovasculature of a wide variety of other solid tumors where it may facilitate endothelial cell sprouting and invasion through its regulation of lytic proteases that have the ability to cleave the extracellular matrix. Similar to the introduction of PSMA-targeting theranostics in prostate carcinoma, overexpression of PSMA on newly formed tumor vessels may serve as a target for imaging and subsequent treatment of cancer through the use of agents that are capable of blocking PSMA in its function or through PSMA-mediated delivery of chemotherapeutics or radiation agents. Preclinical data suggests that PSMA might be involved in cancer-related angiogenesis by degrading the extracellular matrix and participating in integrin signal transduction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed advanced/metastatic solid tumors; any other tumor types documented as PSMA-positive that may benefit from receptor radionuclide therapy and for which there aren't any other effective treatments. For cerebral PSMA-positive tumors, if biopsy is no feasible for technical reasons or risk benefit balance, patients may be enrolled if CT or MRI strongly suggest oncological lesion confirming the 18F- and/or 68Ga PET-CT PSMA positivity;
2. Patients must have measurable disease; patients with prostate cancer who have only bone lesions can be enrolled. See section 9.2 and Appendix D for the evaluation of measurable disease;
3. Relapse or progression of disease on CT/MRI scan and/or WBD-MRI;
4. For patients with prostate cancer: documented radiological progression (in soft tissue and / or bone) and/or biochemical progression (sequence of PSA rising values from a minimal starting value ≥ 1 ng/ml) according to PCWG3;
5. Patients will be admitted to therapeutic phase only if the diagnostic PET/CT PSMA SUV max is ≥ 3;
6. No therapeutic alternatives;
7. Male or Female, aged ≥ 18 years;
8. Life expectancy of greater than 12 weeks;
9. ECOG performance status ≤ 2 (see Appendix A);
10. Patients must have normal organ and marrow function as defined below:

    * leukocytes ≥ 3,000/μL
    * absolute neutrophil count ≥ 1,500/μL
    * haemoglobin ≥ 9 g/dL
    * platelets ≥100,000/μL
    * total bilirubin ≤ 1.5 X institutional upper normal limit (this will not apply to patients with confirmed Gilbert's syndrome)
    * AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional upper normal limit (< 5 X UNL in presence of liver metastases)
    * creatinine ≤ 2 mg/dL
11. A female participant is eligible to participate if she is not pregnant and not breastfeeding. If female of childbearing potential highly effective birth control methods, according to guideline "Recommendation related to contraception and pregnancy testing in clinical trials", (See Appendix F) are mandatory. Highly effective birth control methods are required beginning at the screening visit and continuing until 6 months following last treatment with study drug. Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (1 of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 6 months after final study drug administration. Two acceptable methods of birth control thus include Condom (barrier method of contraception) and one of the following is required ( established use of oral, or injected or implanted hormonal method of contraception by the female partner; placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female partner; additional barrier method like occlusive cap with spermicidal foam/gel/film/cream/suppository in the female partner; tubal ligation in the female partner; vasectomy or other procedure resulting in infertility (eg., bilateral orchiectomy), for more than 6 months;
12. Participant is willing and able to give informed consent for participation in the study.

The participant may not enter the study if ANY of the following apply:

1. Patients who have completed chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) and hormonotherapy within 2 weeks (excluding mCRPC patients), prior to treatment start. A window of 3 days is permitted;
2. All acute toxic effects of any prior therapy (including surgery, radiation therapy, and chemotherapy) must have resolved to a grade ≤ 1 according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE);
3. Participation in another clinical trial with any investigational agents within 30 days prior to study treatment start. A window of 3 days is permitted;
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to 177Lu-PSMAs or other agents used in the study;
5. Medical or psychological conditions that would not allow the participant to understand, or sign the informed consent;
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity rate | 40 months
  safety is evaluated according to version 5.0 of Common Terminology Criteria for Adverse Events (CTCAE). Safety is defined as the percentage of patients who experience acute toxicity grade3/grade4 from the 1st treatment until 30 days after the last treatment cycle.
disease control rate (DCR) | 40 months
  is DCR, defined as the percentage of patients who have achieved complete response, partial response, stable disease (according to RECIST 1.1) or no progression of disease for prostate cancer (according to Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria) at the 1st planned evaluation

SECONDARY OUTCOMES:
progression-free survival (PFS) | 68 months
  PFS is defined as the time from the start treatment date to the date of first observation of documented disease progression (according to RECIST 1.1 or Prostate Cancer Clinical Trials Working Group (PCWG3) criteria for prostate cancer patients) or death due to any cause. Patients without tumor progression at the time of analysis will be censored at their last date of tumor evaluation.
overall survival (OS) | 68 months
  Overall survival is defined as the time from the therapy start to the date of death due to any cause or the date of last contact (censored observation) at the date of data cut-off.
late toxicity | 68 months
  The late toxicity is the toxicity that occurred after 30 days from the last treatment administration up to 6 months.
PET/CT response | 68 months
  PET/CT response is based on Standardized Uptake Value (SUV). PET/CT response will be evaluated with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena Sansovini, MD, Principal Investigator — IRCCS IRST
Locations (2):
- Italy (2):
  - UO Medicina Nucleare, IRCCS IRST, Meldola, Forlì
  - UO Medicina Nucleare, AUSL della Romagna, Cesena

IPD SHARING:
Plan to Share IPD: No